CLINICAL TRIAL: NCT03222856
Title: A Phase II Study of Pembrolizumab and Eribulin in Patients With HR-positive/HER2-negative Metastatic Breast Cancer Previously Treated With Anthracyclines and Taxanes
Brief Title: Ph II Study of Pembrolizumab & Eribulin in Patients With HR+/HER2- MBC Previously Treated With Anthracyclines & Taxanes
Acronym: KELLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP127; 2016-004513-27 (EudraCT Number)
Record Dates: First submitted 2017-07-13; First posted 2017-07-19 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; eribulin

STUDY DESIGN:
Intervention Model Description: A phase II, multicenter, open-label study of pembrolizumab and eribulin in patients with HR- positive/HER2-negative metastatic breast cancer previously treated with anthracyclines and taxanes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + eribulin (Experimental): All eligible patients will be treated with MK3475 (pembrolizumab) 200 mg on day 1 of each 21-day cycle and eribulin 1.23 mg/m2 (equivalent to eribulin mesylate at 1.4 mg/m2) on days 1 and 8 of every 21-day cycle. Treatment with MK3475 (pembrolizumab) and eribulin will continue based on physician criteria. No maximum duration of treatment is specified. Study follow-up will be performed 12 months after last study dose.
  Interventions: Drug: Pembrolizumab; Drug: Eribulin

INTERVENTIONS:
Drug: Pembrolizumab — MK3475 (pembrolizumab) will be supplied directly as a solution for infusion in a single-use vial. Each vial contains 100 mg of MK3475 (pembrolizumab) in 4 ml of solution.
  Other Names: Keytruda; MK3475
Drug: Eribulin — Eribulin will be supplied as a clear and colourless aqueous solution for injection provided in glass vials containing 2 ml. Each 2 ml vial contains eribulin mesylate equivalent to 0.88 mg eribulin.
  Other Names: Halaven

SUMMARY:
This a multicenter, open-label, phase II clinical trial to assess the efficacy of pembrolizumab in combination with eribulin in female patients older than 18 years old with hormone receptor-(HR)positive/HER2-negative metastatic breast cancer (MBC) previously treated with at least one, but not more than two, prior chemotherapeutic regimens for treatment of locally recurrent and/or metastatic disease. Prior therapy must have included an anthracycline and a taxane and prior anti-hormonal therapy is mandatory.

The number of patients to be included is 44 patients at 11 sites. All eligible patients will be treated with MK3475 (pembrolizumab) 200 mg on day 1 of each 21-day cycle and eribulin 1.23 mg/m2 (equivalent to eribulin mesylate at 1.4 mg/m2) on days 1 and 8 of every 21-day cycle.

DETAILED DESCRIPTION:
This a multicenter, open-label, phase II clinical trial to assess the efficacy of pembrolizumab in combination with eribulin in female patients older than 18 years old with hormone receptor-(HR)positive/HER2-negative metastatic breast cancer (MBC) previously treated with at least one, but not more than two, prior chemotherapeutic regimens for treatment of locally recurrent and/or metastatic disease. Prior therapy must have included an anthracycline and a taxane in any combination or order and either in the early or metastatic disease setting unless contraindicated for a given patient. Prior anti-hormonal therapy is mandatory.

The number of patients to be included is 44 patients at 11 sites. The primary objective is to assess the efficacy -as determined by the clinical benefit rate (CBR) (total number of objective responses plus stable disease for at least 24 weeks) based on RECIST v.1.1- of MK3475 (pembrolizumab) in combination with eribulin.

Primary endpoint is CBR based on RECIST v.1.1. All eligible patients will be treated with MK3475 (pembrolizumab) 200 mg on day 1 of each 21-day cycle and eribulin 1.23 mg/m2 (equivalent to eribulin mesylate at 1.4 mg/m2) on days 1 and 8 of every 21-day cycle. Treatment with MK3475 (pembrolizumab) and eribulin will continue based on physician criteria. No maximum duration of treatment is specified. Study follow-up will be performed 12 months after last study dose.

Available tumor tissue for PD-L1 biomarker analysis from a newly obtained core or excisional biopsy since last progression of a metastatic tumor lesion not previously irradiated is requested for this study.

Translational research of this protocol involves the collection, processing, temporary storage, and shipment of samples from consenting patients enrolled in centers selected for participation in the study. The study plan includes collection and initial processing of tumor tissues and blood samples to the central laboratory of Institut Hospital del Mar d"Investigacions Mèdiques (IMIM), that will be used to identify dynamic biomarkers that may be predictive of response to MK3475 (pembrolizumab) and eribulin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures.
2. Female patients ≥18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1 which the Investigator believes is stable at the time of screening.
4. Life expectancy ≥ 12 weeks.
5. Patients have a histologically and/or cytologically confirmed diagnosis of breast cancer.
6. Patients have radiologic evidence of inoperable locally recurrent or MBC.
7. Patients have HER2-negative breast cancer (based on most recently analyzed biopsy) defined as a negative in situ hybridization (ISH) test or an immunohistochemistry (IHC) status of 0, 1+, or 2+ (if IHC 2+, a negative ISH test is required) by local laboratory testing.
8. Patients have HR-positive breast cancer defined as estrogen receptor (ER) and/or progesterone receptor (PR) with >1% of tumor cells positive for ER and/or PR by IHC irrespective of staining intensity.
9. Available tumor tissue for PD-L1 biomarker analysis from a newly obtained core or excisional biopsy since last progression of a metastatic tumor lesion not previously irradiated.

   Note: Subjects for whom tumor biopsies cannot be obtained (e.g., inaccessible tumor or subject safety concern) may submit an archived metastatic tumor specimen only upon agreement from the Sponsor.
10. Patients have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 as assessed by site Investigator and local radiology review.
11. Patients have received at least one, but not more than two, prior chemotherapeutic regimens for locally recurrent and/or metastatic disease. Prior therapy must have included an anthracycline and a taxane in any combination or order and either in the early or metastatic disease setting unless contraindicated for a given patient. Prior anti-hormonal therapy is mandatory.
12. Patients have adequate bone marrow and organ function as defined by the following laboratory values:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
    * Platelets ≥ 100 x 10^9/L.
    * Hemoglobin ≥ 9 g/dL.
    * Potassium, calcium (corrected for serum albumin), and magnesium within normal limits for the institution.
    * Serum creatinine ≤ 1.5 x upper limit of normal (ULN).
    * Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 2.5 x ULN (or ≤ 5.0 x ULN if liver metastases are present).
    * Total serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present). Patients with known Gilbert disease who have serum bilirubin ≤ 3 x ULN may be enrolled.
13. Patients must be accessible for treatment and follow-up.

Exclusion Criteria:

1. Patients have received previous treatment with eribulin and an/or anti-PD1 or anti-PD-L1 agents.
2. Patients have a known hypersensitivity to any of the excipients of MK3475 (pembrolizumab) or eribulin.
3. Patients who have received chemotherapy, targeted small molecule therapy, or radiotherapy within two weeks of first dose of study treatment.
4. Patients who have received monoclonal antibodies for direct antineoplastic treatment or an investigational agent/device within four weeks of first dose of study treatment.
5. Patients have known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

   Note: Known brain metastases are considered active, if any of the following criteria is applicable:
   1. Brain imaging during screening demonstrates progression of existing metastases and/or appearance of new lesions compared to brain imaging performed at least four weeks earlier.
   2. Neurological symptoms attributed to brain metastases have not returned to baseline.
   3. Steroids were used for brain metastases within 28 days of first dose of study treatment.
6. Patients have peripheral neuropathy grade 2 or more.
7. Patients have a concurrent malignancy or malignancy within five years of study enrollment (with the exception of adequately treated, basal or squamous cell skin carcinoma or curatively resected cervical cancer).
8. Patients have not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy.
9. Patients have had a major surgical procedure within 28 days prior to starting study drug.
10. Patients have an active cardiac disease or a history of cardiac dysfunction including any of the following:

    * Unstable angina pectoris or documented myocardial infarction within six months prior to study entry.
    * Symptomatic pericarditis.
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV).
    * Patients have a left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO).
11. Patients have any of the following cardiac conduction abnormalities:

    * Ventricular arrhythmias except for benign premature ventricular contractions.
    * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication.
    * Conduction abnormality requiring a pacemaker.
    * Other cardiac arrhythmia not controlled with medication.
12. Uncontrolled hyper/hypothyroidism or type 1 diabetes mellitus (T1DM). Patients with hypothyroidism stable on hormone replacement will not be excluded from the trial. Patients with controlled T1DM on a stable insulin regimen may be eligible for this study.
13. Active autoimmune disease or a documented history of autoimmune disease, or a syndrome that has required systemic treatment (steroids or immunosuppressive agents) in the past two years.

    Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic steroid replacement therapy (≤ 10 mg prednisone daily) for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Prior allogenic stem cell or solid organ transplantation.
15. Active/history of pneumonitis requiring treatment with steroids or active/history of interstitial lung disease.
16. Active uncontrolled infection at the time of screening
17. Active tuberculosis.
18. Current known infection with HIV.
19. Active hepatitis B (HBV) [patients with negative hepatitis B surface antigen (HBsAg) test and a positive antibody to HBsAg (anti-HBsAg) test at screening are eligible] or hepatitis C (HCV) [patients with a positive antibody to hepatitis C (anti-HCV) are eligible only if polymerase chain reaction (PCR) is negative for virus hepatitis C RNA].
20. Patients have any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment contraindicate patient participation in the clinical study.
21. Treatment with systemic steroids (standard premedication for chemotherapy/contrast reactions, inhaled steroids, and local applications are allowed) or another immunosuppressive agent within seven days prior to study treatment initiation.
22. Has received live vaccines within 30 days prior to first dose of study treatment.
23. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, are not allowed to participate in this study unless they are using highly effective methods of contraception during dosing and up to 120 days after study drugs discontinuation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients age ≥ 18 years with advanced HR-positive/HER2- negative breast cancer previously treated with anthracyclines and taxanes.
Enrollment: 44 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés, PhD, Principal Investigator — MedSIR
Locations (11):
- Spain (11):
  - Corporació Sanitaria Sanitari Parc Taulí, Sabadell, Barcelona
  - Hospital de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital Clínic de Barcelona, Barcelona
  - Instituto Oncológico Baselga - Hospital Quirónsalud Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - MD Anderson, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Garcia JM, Llombart-Cussac A, G Cortes M, Curigliano G, Lopez-Miranda E, Alonso JL, Bermejo B, Calvo L, Caranana V, de la Cruz Sanchez S, M Vazquez R, Prat A, R Borrego M, Sampayo-Cordero M, Segui-Palmer MA, Soberino J, Malfettone A, Schmid P, Cortes J. Pembrolizumab plus eribulin in hormone-receptor-positive, HER2-negative, locally recurrent or metastatic breast cancer (KELLY): An open-label, multicentre, single-arm, phase Ⅱ trial. Eur J Cancer. 2021 May;148:382-394. doi: 10.1016/j.ejca.2021.02.028. Epub 2021 Mar 29. PMID 33794440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Dec 2017 and Oct 2018, a total of 44 patients with HR+ and HER2- MBC were enrolled at 11 sites. These patients were distributed into one arm and treated with pembrolizumab combinated with Eribulin.
Pre-assignment Details: Written informed consent. Females ≥18. ECOG status must be 0 or 1. Life expectancy ≥12 weeks. Patients have histologically and/or cytologically confirmed breast cancer. Radiologic evidence of inoperable lrMBC. HER2-negative breast cancer (by ISH or IHC) of 0,1+,2+. HR-positive BC with >1% of tumor cells. Available tumor tissue for PD-L1 analysis.
Period: Overall Study
Arm/Group | Pembrolizumab + Eribulin
Started | 44
Completed | 37
Not Completed | 7
Not completed — Adverse Event | 6
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 52.50 [46 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 43
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Spain | 44

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Pembrolizumab in Combination With Eribulin.
Description: The efficacy -as determined by the clinical benefit rate (CBR) (total number of objective responses plus stable disease for at least 24 weeks) based on RECIST v.1.1- of MK3475 (pembrolizumab) in combination with eribulin in patients with HR-positive/HER2-negative MBC who have previously received an anthracycline and a taxane (for either early or advanced disease), unless contraindicated, and between one to two lines of chemotherapy in the metastatic setting.
  Per Response Evaluation Criteria In Solid Tumors (RECIST v1.1) for target lesions: Complete Response (CR) is defined as the disappearance of all target lesions. Partial Response (PR) is defined as a decrease of ≥30% in the sum of the longest diameter of target lesions. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as Progressive Disease (PD).
Time Frame: Through study completion. From baseline up to 36 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 44
Participants | 25

2. Secondary Outcome: The CBR in Subjects With Programmed Death Ligand-1 (PD-L1) Positive Tumors.
Description: CBR based on RECIST v.1.1 in subjects with PD-L1 positive tumors.
Time Frame: Through study completion. From baseline up to 36 months.
Population: Patients PD-L1 positive
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 21
Participants | 9

3. Secondary Outcome: The Progression-free Survival (PFS)
Description: PFS based on RECIST v.1.1.
Time Frame: Through study completion. From baseline up to 36 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 44
months | 6.03 [3.7 to 8.4]

4. Secondary Outcome: The PFS in Subjects With PD-L1 Positive Tumors.
Description: PFS based on RECIST v.1.1 in subjects with PD-L1 positive tumors.
Time Frame: Through study completion. From baseline up to 36 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 21
months | 5.27 [2.47 to 6.37]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) represents the time from the start of the study until death from any cause.
Time Frame: From baseline up to 36 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 44
months | 14.23 [9.23 to NA] — The upper limit is reported as Not Available (NA) due to insufficient events or censored data, making accurate estimation unreliable

6. Secondary Outcome: The OS in Subjects With PD-L1 Positive Tumors.
Description: OS in subjects with PD-L1 positive tumors.
Time Frame: Through study completion. From baseline up to 36 months.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 21
months | 13.6 [6.3 to 22.7]

7. Secondary Outcome: Overall Response Rate (ORR) Based on RECIST v1.1
Description: The Overall Response Rate (ORR) is defined as the proportion of participants who achieve a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST v1.1 criteria. ORR is calculated as:
  ORR = (Number of participants with CR + Number of participants with PR) / Total number of participants.
Time Frame: Through study completion. From baseline up to 36 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 44
Participants | 18

8. Secondary Outcome: Overall Response Rate (ORR) in Participants With PD-L1 Positive Tumors Based on RECIST v1.1
Description: The Overall Response Rate (ORR) in participants with PD-L1 positive tumors is defined as the proportion of participants with a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST v1.1 criteria. ORR is calculated as:
  ORR = (Number of participants with CR + Number of participants with PR) / Total number of participants with PD-L1 positive tumors.
Time Frame: Through study completion. From baseline up to 36 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 21
Participants | 8

9. Secondary Outcome: The Duration of Response (DoR)
Description: DoR based on RECIST v.1.1.
Time Frame: Through study completion. From baseline up to 36 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 44
months | 6.23 [3.07 to NA] — There were not enough events in the SOC arm (patients discharged) to estimate the upper limit of the 95% confidence interval.

10. Secondary Outcome: The DoR in Subjects With PD-L1 Positive Tumors.
Description: DoR based on RECIST v.1.1 in subjects with PD-L1 positive tumors.
Time Frame: Through study completion. From baseline up to 36 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 21
months | 5.23 [3.07 to NA] — There were not enough events in the SOC arm (patients discharged) to estimate the upper limit of the 95% confidence interval.

11. Secondary Outcome: Number of AEs Per CTCAE Grade (Safety and Tolerability of Pembrolizumab in Combination With Eribulin)
Description: The safety and tolerability of MK3475 (pembrolizumab) in combination with eribulin according to the US National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.3.
Time Frame: Through study completion. From baseline up to 36 months.
Measure: Number; unit: number of AEs per CTCAE grade
Arm/Group | Pembrolizumab + Eribulin
Number analyzed (Participants) | 44
number of AEs per CTCAE grade
  Grade 1 | 424
  Grade 2 | 192
  Grade 3 | 50
  Grade 4 | 5

12. Other Pre Specified Outcome: Gene Signature Predictive of MK3475 (Pembrolizumab) and Eribulin Therapy Benefit.
Description: New predictive factors of response to MK3475 (pembrolizumab) and eribulin
Time Frame: 24 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: The Link Between Mutational Load and Response to MK3475 (Pembrolizumab) and Eribulin.
Description: New predictive factors of response to MK3475 (pembrolizumab) and eribulin
Time Frame: 24 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: PD-L1 Expression in Circulating Tumor Cells (CTCs) and Its Correlation With Response to MK3475 (Pembrolizumab) and Eribulin.
Description: New predictive factors of response to MK3475 (pembrolizumab) and eribulin
Time Frame: Through study completion. From baseline up to 36 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Safety and tolerability of all patients will be closely monitored throughout study treatment and the follow-up period using the NCI CTCAE v.4.0.3 (36 months)
Arm/Group | Pembrolizumab + Eribulin
All-Cause Mortality (participants affected / at risk) | 11/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 44/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Eribulin (N=44)
Neutropenia (Blood and lymphatic system disorders) | 20 (46)
Anaemia (Blood and lymphatic system disorders) | 19 (32)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (26)
Asthenia (General disorders) | 19 (38)
Diarrhoea (Gastrointestinal disorders) | 14 (30)
Fatigue (General disorders) | 14 (27)
Peripheral neuropathy (Nervous system disorders) | 12 (22)
Nausea (Gastrointestinal disorders) | 11 (18)
Upper respiratory tract infection (Infections and infestations) | 10 (10)
Aspartate aminotransferase increased (Investigations) | 9 (10)
Constipation (Gastrointestinal disorders) | 9 (9)
Mucositis (General disorders) | 9 (17)
Urinary tract infection (Infections and infestations) | 9 (18)
Alanine aminotransferase increased (Investigations) | 8 (14)
Headache (Nervous system disorders) | 8 (12)
Decreased appetite (Metabolism and nutrition disorders) | 7 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Pyrexia (General disorders) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Hypothyroidism (Endocrine disorders) | 5 (6)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Vomiting (Gastrointestinal disorders) | 5 (10)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Blood albumin decreased (Investigations) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Brochitis (Infections and infestations) | 2 (2)
Dizziness (Nervous system disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 4 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Gamma-glutamyltransferase increased (Investigations) | 4 (5)
Groin pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Lacrimation increased (Eye disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Nasopharyngitis (Infections and infestations) | 4 (6)
Platelet count decreased (Investigations) | 3 (3)

LIMITATIONS AND CAVEATS:
There were not enough events in the SOC arm (patients discharged) to estimate the upper limit of the 95% confidence interval in the Duration of Response (DoR) endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03222856/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT03222856/SAP_001.pdf